CLINICAL TRIAL: NCT02897596
Title: Efficacy of GZR/EBR in Early Chronic Hepatitis C in HIV/HCV Co-infected Patients
Acronym: EARLY-HEP-C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARLY-HEP-C
Record Dates: First submitted 2016-08-22; First posted 2016-09-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype 1b (Experimental): Grazoprevir 100 mg/d during 8 weeks. Elbasvir 50 mg/d during 8 weeks.
  Interventions: Drug: Grazoprevir 100 mg/d 8 weeks; Drug: Elbasvir 50 mg/d 8 weeks
- Genotype 1a and 4 (Experimental): Grazoprevir 100 mg/d during 12 weeks. Elbasvir 50 mg/d during 12 weeks.
  Interventions: Drug: Grazoprevir 100 mg/d 12 weeks; Drug: Elbasvir 50 mg/d 12 weeks

INTERVENTIONS:
Drug: Grazoprevir 100 mg/d 8 weeks — Patients with 1b HCV genotype will be received treatment with Grazoprevir (100 mg) during 8 weeks.
  Other Names: MK-5172 100 mg
  Arms: Genotype 1b
Drug: Elbasvir 50 mg/d 8 weeks — Patients with 1b HCV genotype will be received treatment with Elbasvir (50mg) during 8 weeks.
  Other Names: MK-8742 50 mg
  Arms: Genotype 1b
Drug: Grazoprevir 100 mg/d 12 weeks — Patients with 1a or 4 HCV genotype will be received treatment with Grazoprevir (100 mg) during 12 weeks.
  Other Names: MK-5172 100 mg
  Arms: Genotype 1a and 4
Drug: Elbasvir 50 mg/d 12 weeks — Patients with 1a or 4 HCV genotype will be received treatment with Elbasvir (50mg) during 12 weeks.
  Other Names: MK-8742 50 mg
  Arms: Genotype 1a and 4

SUMMARY:
Evaluate the efficacy of 12 or 8 weeks treatment with Grazoprevir/Elbasvir in Early Chronic Hepatitis C GT1,4 in HIV co-infected patients and evaluate the safety and tolerability of Grazoprevir + Elbasvir in HIV-HCV co-infected patients.

DETAILED DESCRIPTION:
Genotype 1b: 8 weeks treatment with Grazoprevir/Elbasvir

Genotype 1a and 4: 12 weeks treatment with Grazoprevir/Elbasvir

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Patients with early chronic hepatitis C (Genotype 1 or 4) which is defined as chronic hepatitis C with known episode of AHC within the last 4 years including those who failed to PEG/RBV or those who never received therapy for AHC. AHC infection is diagnosed on the basis of documented HCV-RNA positivity (> 10.000 IU/mL) and anti-HCV seroconversion.
* No history of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs/symptoms of advanced liver disease
* Have liver disease staging assessment as follows: Fibroscan performed within 3 previous months of Day 1 of this study showing result <8 kPa
* Be HIV-1 infected, documented by any licensed rapid HIV test and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load.
* Be on stable HIV Antiretroviral Therapy (ART) for at least 8 weeks prior to study entry using a dual NRTI backbone of tenofovir or abacavir

Exclusion Criteria:

* < 18 years of age
* Patients with chronic hepatitis C genotypes other than 1 or 4.
* History of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs/symptoms of advanced liver disease
* Have liver disease staging assessment as follows: Fibroscan performed within 3 previous months of Day 1 of this study showing result > 8kPa
* Not be HIV-1 infected, documented by any licensed rapid HIV test and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load.
* Due to known or suspected drug-drug interactions, for the purpose of this study, the use of Non Nucleoside Reverse Transcriptase Inhibitors, Inhibitors or Protease Inhibitors against HIV will be not allow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-04-28 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response. | 24 weeks
  Sustained virological response 12 (SVR12) defined as HCV-RNA undetectable at post-treatment.

SECONDARY OUTCOMES:
Reinfection rate | 1 year
  Evaluate the reinfection rate during 1 year of follow-up Sustained virological response defined as HCV-RNA undetectable at post-treatment.
Evaluate the safety and tolerability by means of number of participants with treatment-related adverse events. | 2 years
  number of adverse events treatment-related assess in 62 patients.
Evaluate the emergence of of viral resistance-associated variants (RAV) resistant to MK-5172 and MK-8742. during the follow up. | 2 years
  In case of viral failure confirmation during the follow up, viral resistence-associated variants will be assess by samples genotyping HCV protease and NS5A gene at baseline and after the viral failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico y provincial de Barcelona, Barcelona, Spain